CLINICAL TRIAL: NCT07024251
Title: BIOlogical Waste Sample Collection for Progress in Oral and MAXillofacial Research
Acronym: BIO-MAX
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-MAX
Record Dates: First submitted 2025-05-19; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Oral and Maxillofacial Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The study collects saliva (mandatory), crevicular fluid, gingival tissue, teeth, bone fragments, adipose tissue, blood, and intra-cystic fluid for analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing routine oral exams or elective oral and maxillofacial surgery.: Adult male and female patients (18+) undergoing oral exams or elective oral/maxillofacial surgery at IRCCS Galeazzi.

SUMMARY:
The BIO-MAX (BIOlogical waste sample collection for progress in oral and MAXillofacial research) study, led by IRCCS Ospedale Galeazzi-Sant'Ambrogio, is a five-year observational research project aimed at improving the understanding and treatment of oral and maxillofacial conditions.

Researchers are collecting and analyzing biological samples-such as saliva, blood, and tissues typically discarded during dental and surgical procedures-from adult patients visiting the hospital for oral exams or surgery. A key focus is the study of salivary irisin, a promising biomarker linked to diseases like diabetes and heart disease. By examining how irisin levels vary with age, gender, lifestyle, and oral health, the team hopes to establish baseline values and better understand its diagnostic potential.

In addition to irisin analysis, the study will explore other waste tissues to uncover disease mechanisms, identify new biomarkers, and test future therapies using patient-derived laboratory models. Overall, BIO-MAX seeks to enhance diagnostics, improve patient care, and pave the way for innovative treatments in oral and maxillofacial medicine.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* ≥18 years old
* patients undergoing either routine oral clinical examination or elective oral and maxillofacial surgery at IRCCS Ospedale Galeazzi - Sant'Ambrogio

Exclusion Criteria:

* <18 years old
* inability to sign the Informed Consent
* positivity to virological tests (HIV, HCV, HBV, TPHA), if serological analysis is required
* pregnancy and breast feeding with declaration of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After informed consent, eligible patients undergoing routine exams or elective oral and maxillofacial surgery will be enrolled for biological waste collection.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Salivary Irisin Concentration Measured by Enzyme-Linked Immunosorbent Assay (ELISA) | 5 years from first patient enrollment
  Description:
  Salivary irisin concentration will be measured in all participants using a validated enzyme-linked immunosorbent assay (ELISA). Measurements will be reported in ng/mL, aiming to provide a comprehensive profile of salivary irisin levels in relation to demographic, lifestyle, medical, and health-related variables.
  Additional details:
  Irisin concentration data will be analyzed in relation to participant characteristics such as age (in years), gender, physical activity level, body mass index (BMI in kg/m²), oral health status (assessed through clinical dental examination), self-reported general health status, and current pharmacological treatments. These variables will serve as contextual covariates to explore associations and subgroup differences in irisin levels. Although some covariates involve quantitative measurements, they are not considered outcome measures and will be used solely to support interpretation of the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No